CLINICAL TRIAL: NCT02744612
Title: A Multi-Center Phase II Trial of Ibrutinib Plus Brentuximab Vedotin in Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Ibrutinib and Brentuximab Vedotin in Treating Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15334; NCI-2016-00176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15334 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-02-22; First posted 2016-04-20 (Estimated); Results first posted 2023-07-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 days (Experimental): Patients receive ibrutinib 420 mg PO QD on days 1-21 and brentuximab vedotin 1.8 mg/kg IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Ibrutinib
- Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 days (Experimental): Patients receive ibrutinib 560 mg PO QD on days 1-21 and brentuximab vedotin 1.8 mg/kg IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Drug: Ibrutinib

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765

SUMMARY:
This phase II trial studies how well ibrutinib and brentuximab vedotin work in treating patients with Hodgkin lymphoma that has returned (relapsed) or does not respond to treatment (refractory). Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as brentuximab vedotin, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving ibrutinib together with brentuximab vedotin may be a better treatment for Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the anti-tumor activity of the two agent combination ibrutinib and brentuximab vedotin, as assessed by complete response (CR) rate.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of the two agent combination through evaluation of toxicities, including type, frequency, severity, attribution, time course and duration.

II. Obtain estimates of overall response rate (ORR), response duration and survival (overall and progression-free).

III. Describe outcomes of patients who ultimately undergo autologous or allogeneic hematopoietic cell transplantation following treatment with ibrutinib/brentuximab vedotin.

EXPLORATORY OBJECTIVE:

I. Collect deoxyribonucleic acid (DNA)/ribonucleic acid (RNA) from lymphoma specimens and serial plasma samples for future biomarker evaluation.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-21 and brentuximab vedotin intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented or cytologically confirmed Hodgkin lymphoma with CD30 expression
* Patients must have absolute neutrophil count (ANC) >= 1000/uL; neupogen can be given before and during treatment to achieve target ANC >= 1000/uL
* Patients must have platelets (plt) >= 50,000/uL; platelet transfusion and packed red blood cell transfusion can also be given prior to the start of treatment and during treatment to achieve a target plt >= 50,000/uL provided that patients have not received growth factors for at least 14 days prior to entering trial
* Patients must have hemoglobin >= 8.5 g/dl; platelet transfusion and packed red blood cell transfusion can also be given prior to the start of treatment and during treatment to achieve a target hemoglobin of >= 8.5/ul provided that patients have not received growth factors for at least 14 days prior to entering trial
* Patients must have measurable disease > 1.5 cm evidenced by computed tomography (CT) scan of the neck/chest/abdomen (abd)/pelvis or CT/positron emission tomography (PET) scans
* Patients must be either refractory to or relapsed after 1 line of therapy
* Prior radiation therapy is allowed
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method of contraception for the duration of the study
* Over 40 kg; life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) of 0-2
* Total bilirubin within 1.5 x the upper limit of normal institutional limits; patients with elevation of unconjugated bilirubin alone, as in Gilbert's disease, are eligible
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal (unless demonstrated Hodgkin lymphoma involvement of the liver); estimated creatinine clearance >= 30 ml/min (Cockcroft-Gault) and/or 24 urine analysis as needed
* Prothrombin time (PT)/international normalized ratio (INR) < 1.5 x upper limit of normal (ULN) and partial thromboplastin time (PTT) (activated PTT [aPTT]) < 1.5 x ULN
* The effects of brentuximab vedotin and ibrutinib on the developing fetus is unknowm; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent; they are to give voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Patient must be either refractory to or relapsed after 1 line of therapy
* Prior hematopoietic transplantation is allowed (autologous and/or allogeneic)
* Prior brentuximab vedotin is allowed provided that patients were not refractory (defined as developing progressive disease while on treatment or progressed within 3 months of finished last dose of brentuximab vedotin)
* Prior ibrutinib for Hodgkin lymphoma is not allowed

Exclusion Criteria:

* Less than or equal to 40 kg
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological therapy, chemotherapy, or radiation therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib and brentuximab vedotin (BV)
* Patients must not have received prior chemotherapy or radiation for =< 3 weeks before study enrollment, or those who have not recovered from the adverse events due to agents administered more than 3 weeks earlier are excluded
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Significant screening electrocardiogram (ECG) abnormalities including, but not limited to, left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) >= 470 msec; subjects with a cardiac pacemaker who have a QTc interval of >= 470 msec may be eligible if these findings are considered not clinically significant as documented via a cardiology evaluation
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients with active central nervous system (CNS) disease or history of brain metastases are excluded from study
* Patients may be on steroids prior to initiation of treatment, provided that, by cycle 1 day 1, steroids use was tapered down to less than or equal to 20 mg of prednisone
* Pregnant women are excluded from this study because of the potential teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent infection requiring systemic treatment that was completed =< 14 days before the first dose of study drug
* Known active infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV); testing to be done only if patients suspected of having infections or exposures; subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded; subjects who have an undetectable human immunodeficiency virus (HIV) viral load with CD4 >= 200 and are on highly active antiretroviral therapy (HAART) medication are allowed
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* STUDY-SPECIFIC EXCLUSIONS:
* Patient has hypersensitivity to brentuximab vedotin
* Refractory to prior brentuximab vedotin (defined as developing progressive disease while on treatment or progressed within 3 month of finished last dose of brentuximab vedotin)
* No active graft-versus-host disease (GVHD) or on immunosuppressive medication for GVHD
* Recent infection requiring intravenous anti-infective treatment that was completed =< 14 days before the first dose of study drug
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), grade 0 or 1, or to the levels dictated in the inclusion/exclusion criteria, with the exception of alopecia
* Baseline grade II peripheral neuropathy
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Major surgery within 4 weeks of first dose of study drug
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Herrera, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days
Started | 3 | 36
Completed | 3 | 34
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Total
Number analyzed (Participants) | 3 | 36 | 39
Age, Continuous [Median (Full Range); unit: years] | 34 [21 to 52] | 33 [17 to 71] | 33 [17 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 1 | 25 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 16 | 16
  Not Hispanic or Latino | 3 | 18 | 21
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 36 | 39

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Complete response is defined based on Cheson criteria [Cheson BD, Fisher RI, Barrington SF, et al: Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification. Journal of Clinical Oncology 32:3059-3067, 2014]. The complete response rate was calculated as the percent of evaluable patients that have confirmed CR; exact 95% confidence intervals was calculated for this estimate.
Time Frame: Up to 8 months.
Population: 3 subjects didn't complete Cycle 1 and then were off treatment. So they are not evaluable for response.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days
Number analyzed (Participants) | 3 | 33
percent of participants | 0 [0 to 71] | 36 [20 to 55]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The overall response rate was calculated as the percent of evaluable patients that have confirmed complete response (CR) or partial response (PR); exact 95% confidence intervals will be calculated for this estimate. CR and PR are defined based on Cheson criteria [Cheson BD, Fisher RI, Barrington SF, et al: Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification. Journal of Clinical Oncology 32:3059-3067, 2014].
Time Frame: Up to 8 months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days
Number analyzed (Participants) | 3 | 33
percent of participants | 33 [1 to 91] | 67 [48 to 82]

ADVERSE EVENTS:
Time Frame: From the time of the first study treatment up to 2 years post treatment, an average of 28 months.
Arm/Group | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/36
Serious Adverse Events (participants affected / at risk) | 0/3 | 10/36
Other Adverse Events (participants affected / at risk) | 3/3 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days (N=3) | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Ibrutinib 420 mg PO QD + BV 1.8 mg/kg IV Q21 Days (N=3) | Arm II: Ibrutinib 560 mg PO QD + BV 1.8 mg/kg IV Q21 Days (N=36)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 15 (29)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 2 (5)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 6 (11)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (4)
Abdominal distension (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Ear and labyrinth disorders) | 0 (0) | 13 (17)
Bloating (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Colitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Ear and labyrinth disorders) | 0 (0) | 13 (15)
Diarrhea (Ear and labyrinth disorders) | 1 (1) | 23 (38)
Dry mouth (Ear and labyrinth disorders) | 0 (0) | 7 (7)
Dyspepsia (Ear and labyrinth disorders) | 0 (0) | 10 (13)
Dysphagia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Flatulence (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastritis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Ear and labyrinth disorders) | 1 (1) | 5 (5)
Gastrointestinal disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 9 (16)
Gastrointestinal pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ileus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Mucositis oral (Ear and labyrinth disorders) | 0 (0) | 5 (7)
Nausea (Ear and labyrinth disorders) | 2 (2) | 25 (42)
Oral pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Stomach pain (Ear and labyrinth disorders) | 1 (1) | 5 (9)
Vomiting (Ear and labyrinth disorders) | 1 (2) | 15 (26)
Chills (General disorders) | 0 (0) | 9 (9)
Edema face (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 5 (5)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 19 (34)
Fever (General disorders) | 2 (2) | 14 (15)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 4 (7)
Infusion related reaction (General disorders) | 0 (0) | 7 (13)
Localized edema (General disorders) | 0 (0) | 4 (4)
Malaise (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 6 (8)
Pain (General disorders) | 0 (0) | 7 (8)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 6 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 16 (24)
Alkaline phosphatase increased (Investigations) | 1 (1) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 13 (18)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (4)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 8 (11)
Neutrophil count decreased (Investigations) | 0 (0) | 10 (21)
Platelet count decreased (Investigations) | 1 (1) | 17 (25)
Weight gain (Investigations) | 0 (0) | 1 (3)
Weight loss (Investigations) | 0 (0) | 2 (3)
White blood cell decreased (Investigations) | 0 (0) | 9 (18)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 13 (17)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 9 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 7 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 10 (16)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 13 (23)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 6 (9)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 13 (18)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 11 (13)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (13)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (11)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 11 (20)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 17 (29)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 22 (48)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 6 (8)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 9 (16)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 6 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 8 (9)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (4)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 10 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (15)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 15 (31)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 16 (38)
Hypotension (Vascular disorders) | 2 (2) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT02744612/Prot_SAP_000.pdf